CLINICAL TRIAL: NCT04504396
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Trial Comparing the Efficacy and Safety of PB-119 in Combination With Metformin in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin Alone
Brief Title: Safety and Efficacy of PB-119 in Subjects With Type 2 Diabetes and Not Well-controlled by Metformin Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB119302
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-119 once-weekly-subcutaneous injection (Experimental): PB119 (polyethylene glycol exenatide) is a long-acting GLP-1RA for injection, which will be administered 150μg once-weekly subcutaneously to patients in active drug group for 24 weeks.
  Interventions: Drug: GLP-1 receptor agonist
- Placebo once-weekly-subcutaneous injection (Placebo Comparator): PB-119 150μg matched placebo which will be used in placebo group for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-1 receptor agonist — PB-119 is an investigational pegylated human glucagon-like peptide-1 (GLP-1) receptor agonist. The dosing regimen is 150μg once every week as subcutaneous administration. Patients in PB-119 group will be administered the active drugs for 52 weeks (24+28).
  Arms: PB-119 once-weekly-subcutaneous injection
Drug: Placebo — PB-119 matched placebo will be used once every week as subcutaneous administration to placebo group for 24 weeks.
  Other Names: PB-119 Placebo
  Arms: Placebo once-weekly-subcutaneous injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of 24 once-weekly subcutaneous doses of PB-119 to subjects with type 2 diabetes mellitus (T2DM) not well-controlled by metformin monotherapy.

DETAILED DESCRIPTION:
This is a phase 3 multicenter, randomized, double-blind, placebo-controlled, parallel dose cohort study to evaluate the efficacy and safety of PB-119 to patients with T2DM not well-controlled by metformin monotherapy. Patients will be assessed for eligibility over a 2 week screening period prior to a 4-week run-in period,a 24-week double-blind treatment period and a 28-week open-label treatment period. The eligible patients will be randomized to PB-119 or placebo cohort at a 1:1 ratio for the first 24-week. Patients in PB-119 group will subsequently be given active drug and patients in placebo group will take placebo, all patients in two groups will remain metformin background therapy. In the 28-week open-label period, all patients will be administered active drugs. After that, there will be a 4-week follow-up period; All randomized patients will be taken blood samples for the pharmacokinetic (PK) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18~75 years old;
* T2DM and treated with Metformin ≥ 1500mg/day or maximum tolerated dose(≥1000mg,<1500mg) constantly for at least 8 consecutive weeks;
* 7.5% ≤ HbA1c ≤ 10.0% at screening;
* 18.5 kg/m2 < BMI < 40.0 kg/m2 at screening;

Exclusion Criteria:

* Any anti-diabetic therapy other than Metformin within 8 weeks before screening；
* T1DM;
* Received insulin therapy more than 14 days within 1 year before screening;
* Female who is pregnant, breast-feeding;
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol;
* History of acute diabetic complications, such as diabetic ketoacidosis or hyperglycemic hyperosmolar status within 6 months before screening；
* History or presence of pancreatitis (acute or chronic);
* Presence or history of malignant neoplasms within the past 5 years prior to the day of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | week 1, week 25
  Change in HbA1c from baseline(week 1) to week 25

SECONDARY OUTCOMES:
HbA1c Below 7.0% | week 1, week 25
  Percentage of participants with HbA1c below 7.0% was evaluated at week 25.
Change in Body Weight (kg) | week 1, week 25
  Change from baseline (week 1) in body weight was evaluated at week 25
Change in Fasting Plasma Glucose (FPG) | week 1, week 25
  Change from baseline (week 1) in FPG was evaluated at week 25
Change in Body Mass Index | week 1, week 25
  Change from baseline (week 1) in body mass index (BMI) was evaluated at week 25.

CONTACTS AND LOCATIONS:
Overall Officials: HuiMin Zhou, MD，PhD, Principal Investigator — First Hospital of Hebei Medical University; WeiHong Song, MD，PhD, Principal Investigator — First People's Hospital of Chenzhou; YanJun Wang, MD，PhD, Principal Investigator — Second Hospital of Jilin University; Jing Yang, MD，PhD, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Bin Gao, MD，PhD, Principal Investigator — Tang-Du Hospital; XinLing Wang, Doctor, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region; MingHui Hou, MD，PhD, Principal Investigator — Affiliated Hospital of Hebei University; Lin Liao, MD，PhD, Principal Investigator — Qianfoshan Hospital; Linong Ji, MD，PhD, Principal Investigator — Beijing University People's Hospital; Minxiu Yao, MD，PhD, Principal Investigator — Qingdao Central Hospital; Huige Shao, MD，PhD, Principal Investigator — Changsha Central Hospital; Jingna Lin, MD，PhD, Principal Investigator — Tianjin People's Hospital; Xiaohong Lin, MD，PhD, Principal Investigator — ZhuZhou Central Hospital; Jianhua Ma, MD，PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Wei Zhang, MD，PhD, Principal Investigator — Qiqihar First Hospital; Hui Liu, MD，PhD, Principal Investigator — Luoyang Central Hospital; Tao Ning, MD，PhD, Principal Investigator — Baotou Central Hospital; Xiaohong Wu, MD，PhD, Principal Investigator — Zhejiang Province People's Hospital; Xueying Wang, MD，PhD, Principal Investigator — Jingzhou Central Hospital; Lan Xu, MD，PhD, Principal Investigator — WuXi Central Hospital
Locations (1):
- Beijing University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No